CLINICAL TRIAL: NCT06715423
Title: High Flow Nasal Oxygen Therapy an Implementation Study in Pediatric Wards
Acronym: HFNO
Status: Not yet recruiting | Type: Observational
Sponsor: Epicentre (Other)
Collaborators: MOH Afghanistan (Unknown); MOH Bangladesh (Unknown); MOH Sierra Leone (Unknown); MOH Yemen (Unknown); MSF Médecins Sans Frontières Belgium (Unknown); MSF Médecins Sans Frontières France (Unknown); Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: G2429-HFNO_ProcessEvaluation
Record Dates: First submitted 2024-11-26; First posted 2024-12-04 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Moderate Respiratory Distress; Severe Respiratory Distress
Keywords: oxygen; high flow; pneumonia; pediatrics
MeSH Terms: conditions — Dyspnea; Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediactric ICU Hospitalized children 1mo to 5 yo: Prescription of HFNO therapy

SUMMARY:
The purpose of this study is to prospectively evaluate the process of implementing HFNO in several MSF projects, varying according to geographical and programmatic contexts, population, health structures, human resources, and management. It will generate evidence on the operational feasibility (in terms of human resources, equipment, logistics and costs) of integrating HFNO into PICU standard of care, as well as on the users' and caregivers' perspectives on HFNO and on the children clinical outcomes observed where HFNO is implemented. This relevant information will guide MSF in the decision making of scaling up HFNO therapy in its projects.

DETAILED DESCRIPTION:
Mixed method study: quantitative component for the data of the children and qualitative data for the perception for health staffs and parents

ELIGIBILITY:
Inclusion Criteria:

* prescription of HFNO by clinician
* parent consenting to the use of the data

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: MSF pediatric ICU in 4 sites (Herat- Afghanistan, Kenema- Sierra Leone, Goyalmara hospital for Rohingya refugee - Bangladesh, Khamir- Yemen)
Sampling Method: Non-Probability Sample
Enrollment: 960 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Recovery with SPO2 above 92% | From enrollment to day 3 to 10

OTHER OUTCOMES:
Acceptability, feasibility and perception from the caretaker point of view | 2 weeks after hospitalisation
  interview of the caretaker
Acceptability, feasibility and perception from the health staff point of view | From Month 2 until Month 12
  Interview of the health staffs (doctors, nurses, biomed, managers, logisticians)

CONTACTS AND LOCATIONS:
Locations (1):
- Herat regional Hospital, Herat, Afghanistan

IPD SHARING:
Plan to Share IPD: Yes
Based on the data sharing policy of MSF
Supporting Information: CSR